CLINICAL TRIAL: NCT02726087
Title: Health-related Quality of Life, Satisfaction and Outcomes After Ministernotomy Versus Full Sternotomy Aortic Valve Replacement. A Randomized Controlled Trial (QUALITY-AVR TRIAL)
Brief Title: Quality of Life After Ministernotomy Versus Full Sternotomy Aortic Valve Replacement
Acronym: QUALITY-AVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Principal Investigator, Emiliano Rodriguez-Caulo, MD, PhD, FETCS, Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CALIDAD-SVAO
Record Dates: First submitted 2016-03-13; First posted 2016-04-01 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases; Aortic Valve Disease
Keywords: Ministernotomy; aortic valve stenosis; quality of life; satisfaction; cardiac surgery
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Aortic Valve Disease; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ministernotomy (Experimental): Minimally invasive aortic valve replacement with Partial "J" upper hemisternotomy through right 4th intercostal space, performed according to current standard of care practice.
  Interventions: Procedure: ministernotomy
- full sternotomy (Active Comparator): Full sternotomy AVR through a standard median sternotomy, performed according to current standard of care practice.
  Interventions: Procedure: Full sternotomy

INTERVENTIONS:
Procedure: ministernotomy — Partial upper "J" hemisternotomy trough 4th right intercostal space)
  Arms: ministernotomy
Procedure: Full sternotomy — Conventional full median sternotomy
  Arms: full sternotomy

SUMMARY:
This is a single-center, single-blind, all comer, randomized controlled trial. Patients scheduled for isolated aortic valve replacement (AVR) due to aortic stenosis at "Virgen de la Victoria Universitary Hospital", Málaga, Spain, will be eligible. Ninety-six patients will be randomly assigned to either partial upper sternotomy (ministernotomy, 48 patients) or full sternotomy AVR (48 patients). Sample size was determined for an Alpha error of 0.05,and Beta error of 0.1 for a power of 90% in detecting 0.10 difference points in quality of life EQ-5D-5L-index or 10 points in EQ-5D-5L-Visual Analogic Scale (QOL).

DETAILED DESCRIPTION:
This is a single-center, single-blind, all comer, randomized controlled trial. Patients scheduled for isolated aortic valve replacement (AVR) due to aortic stenosis at "Virgen de la Victoria Universitary Hospital", Málaga, Spain, will be eligible. Ninety-six patients will be randomly assigned to either partial upper sternotomy (ministernotomy, 48 patients) or full sternotomy AVR (48 patients). Sample size was determined for an Alpha error of 0.05,and Beta error of 0.1 for a power of 90% in detecting 0.10 difference points in quality of life EQ-5D-5L-index or 10 points in EQ-5D-5L-Visual Analogic Scale.

Inclusion criteria is severe aortic stenosis referred for medically indicated isolated aortic valve replacement due to aortic stenosis in patients >18 years.

Exclusion criteria are left ventricular ejection fraction less than 40%, previous cardiac surgery, urgent/emergent surgery, infective endocarditis, need of concomitant procedures other than isolated Morrow miectomy and thorax deformity.

CE-marked and FDA-approved mechanical (Sorin Carbomedics®) and stented bioprosthetic aortic valves will be implanted (Carpentier Edwards Perimount® and Sorin Crown®). Perceval S Sutureless bioprosthetic valves (LivaNova®) could be used if needed in very small aortic annulus or high risk patients Quality of Life postoperative outcomes will be assessed, as QOL measurements and health status with the EQ-5D-5L® questionnaire (QOL index, health visual analogic scale, severity index and health index), repeatedly assessed preoperatively and postoperatively at 1-6-12 months. Clinical postoperative complications and outcomes will be registered at 1 month and 1 year as main secondary and safety end-point (combined end-point of 4 and 6 major complications) Patient Satisfaction will be assessed with a 20 question cardiac-surgery specific satisfaction questionnaire (SATISCORE®).

Survival will be assessed at 1 year. Clinical pre and postoperative characteristics will be registered. Routine blood sampling will be performed pre- and postoperatively. All available data will be collected prospectively. Informed consent) will be obtained from patients meeting the inclusion criteria before the initiation of any study-specific procedures.

The Institutional Review Board Ethic Comittee approved this study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Severe aortic stenosis defined as aortic valve area of less than 1 cm2 or index area of 0.6 cm2/m2 or mean gradient greater than 40 mmHg by echocardiography or double lesion with predominant stenosis.
* Referred for medically indicated aortic valve replacement
* Provide written informed consent

Exclusion Criteria:

* Left ventricular ejection fraction less than 0.40
* Presence of any coexisting severe valvular disorder
* Previous cardiac surgery
* Urgent or emergent surgery
* Infective endocarditis
* Need for concomitant procedures other than isolated myectomy
* Severe COPD
* Severe thorax deformity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-03-20; Primary Completion 2019-05-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
Differences between intervention groups in change from baseline Questionnaire EQ-5D-5L® Index at 1, 6 or 12 months | baseline-1-6-12 months
  Questionnaire EQ-5D-5L® for quality of life

SECONDARY OUTCOMES:
Differences between intervention groups in change from baseline Questionnaire EQ-5D-5L® Visual Analogic Scale for pain at 1, 6 or 12 months | baseline-1-6-12 months
  Questionnaire EQ-5D-5L® for quality of life
Early postoperative combined endpoint of 6 complications | 1 month
  All cause Mortality, acute myocardial infarction, cerebrovascular or transient ischemic accident, acute renal failure AKIN (acute kidney injury classification) greater or equal than 2, nosocomial infections (Pneumonia, early endocarditis, mediastinitis, sepsis) and need of any reintervention
Satiscore Questionnaire | 1-6 months
  Satisfaction in cardiac surgery
Differences between intervention groups in change from baseline Questionnaire EQ-5D-5L® severity index at 1, 6 and 12 months | baseline-1-6-12 months
  Questionnaire EQ-5D-5L® for quality of life
Differences between intervention groups in change from baseline Questionnaire EQ-5D-5L® health index (severity index inverse) at 1, 6 and 12 months | baseline-1-6-12 months
  Questionnaire EQ-5D-5L® for quality of life
Late postoperative combined endpoint of 6 complications | 1-5 years
  All cause Mortality, acute myocardial infarction, cerebrovascular or transient ischemic accident, acute renal failure AKIN (acute kidney injury classification) greater or equal than 2, nosocomial infections (Pneumonia, early endocarditis, mediastinitis, sepsis) and need of any reintervention
Total in-Hospital and Intensive Care Unit stay (in days) | From date of surgery until the date of discharge or date of death from any cause, whichever came first, assessed up to 1 year
Cardiopulmonary bypass time in minutes and cross-clamp ischemic heart time in minutes needed in the surgery | day 1 after surgery
Mechanical Ventilatory Support time needed after surgery (in hours) | 7 days
Transfusional requirements (number of red packed cells, fresh frozen plasma and platelets) | First 72 hours after surgery
New York Heart Association functional class scale for heart failure | baseline-1-6-12 months
  To assess heart failure status between participants
Number of participants alive (Survival) | 6-12 months
  To assess first year mortality
Number of participants alive (Survival) | 5 years
  To assess 5 year mortality
Early postoperative combined endpoint of 4 complications | 1 month
  All cause Mortality, acute myocardial infarction, cerebrovascular or transient ischemic accident, and acute renal failure AKIN (acute kidney injury classification) greater or equal than 2,
Late postoperative combined endpoint of 4 complications | 1-5 years year
  All cause Mortality, acute myocardial infarction, cerebrovascular or transient ischemic accident, and acute renal failure AKIN (acute kidney injury classification) greater or equal than 2,

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano A Rodriguez-Caulo, MD,PhD,FECTS, Principal Investigator — Hospital Universitario Virgen de la Victoria, Málaga, spain
Locations (1):
- Hospital Universitario Virgen de La Victoria, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Caulo EA, Guijarro-Contreras A, Otero-Forero J, Mataro MJ, Sanchez-Espin G, Guzon A, Porras C, Such M, Ordonez A, Melero-Tejedor JM, Jimenez-Navarro M. Quality of life, satisfaction and outcomes after ministernotomy versus full sternotomy isolated aortic valve replacement (QUALITY-AVR): study protocol for a randomised controlled trial. Trials. 2018 Feb 17;19(1):114. doi: 10.1186/s13063-018-2486-x. PMID 29454380